CLINICAL TRIAL: NCT06383637
Title: Assessment of Knowledge, Attitude and Practice (KAP) Regarding Antibiotics and Antibiotic Resistance Among Dental Interns: Multicenter Cross Sectional Study
Brief Title: Antibiotic Use and Resistance KAP Among Dental Interns
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Attia, Lecturer, Cairo University
Other Study IDs: KAP-ABR-Interns
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic Side Effect; Antibiotic Resistant Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is designed as a cross-sectional online-based questionnaire, and it will be distributed among dental interns. Assess the following among dental interns (1) The knowledge, attitude, and practices (KAP) towards antibiotics and antibiotic resistance; (2) The correlation between their KAP score and where they spend their internship year? (4) Development of the curriculum to provide sufficient training and information about antibiotics and antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Dental interns

Exclusion Criteria:

* undergraduates dental students
* postgraduates dental students

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: dental interns
Sampling Method: Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge of dental interns regarding antibiotic use and resistance | 6 Months
  KAP questionnaire

IPD SHARING:
Plan to Share IPD: Undecided